CLINICAL TRIAL: NCT05107336
Title: A Randomised, Single-Blind, Placebo-Controlled, Phase I Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD2693 Following Multiple Subcutaneous Dose Administration in Healthy Participants
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics (Movement of Drugs Within the Body) of AZD2693 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: D7830C00006
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetics; Healthy Japanese Participants; Non-alcoholic fatty liver disease; Non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study center staff including the Investigator have to remain blinded during the clinical conduct of a given cohort with regard to study intervention (AZD2693 or placebo). The study will be blinded for all study personnel including the Investigator during the clinical conduct of the study and the Sponsor will remain blinded up to the unblinded safety review committee review of the data from the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1: AZD2693 (Experimental): Japanese Participants will receive Dose A of AZD2693.
  Interventions: Drug: AZD2693
- Cohort 2: AZD2693 (Experimental): Japanese Participants will receive Dose B of AZD2693.
  Interventions: Drug: AZD2693
- Cohort 3: AZD2693 (Experimental): Japanese Participants will receive Dose C of AZD2693.
  Interventions: Drug: AZD2693
- Cohort 4: AZD2693 (Experimental): Non-Asian Participants will receive Dose C of AZD2693
  Interventions: Drug: AZD2693
- Placebo (Placebo Comparator): Japanese and Non-Asian Participants will receive placebo matching Dose A, B, and C to AZD2693.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2693 — Participants will receive subcutaneous injection of AZD2693, once per month.
  Arms: Cohort 1: AZD2693; Cohort 2: AZD2693; Cohort 3: AZD2693; Cohort 4: AZD2693
Drug: Placebo — Participants will receive subcutaneous injection of placebo (volume matching to AZD2693 injection [0.9% saline solution]), once per month.
  Arms: Placebo

SUMMARY:
This Phase I, randomised, single-blind, placebo-controlled study has been designed to assess the safety, tolerability, and pharmacokinetics (PK) of AZD2693 following subcutaneous (SC) administration of AZD2693 in healthy participants

DETAILED DESCRIPTION:
The study will be performed at a single study center in Japan.

The study will comprise of following periods:

* Screening Period of maximum 28 days.
* An 8-week Treatment Period during which participants will be randomized to receive multiple doses of AZD2693 or placebo at the study center.
* A Follow-up Period of 15 weeks post last dose of study intervention consisting of 8 Follow-up Visits.

Participants will be enrolled in 4 consecutive cohorts of 11 participants where 8 participants will be randomized to receive AZD2693 and 3 participants will be randomized to receive placebo.

A participant is considered to have completed the study if the participant has completed all phases of the study including the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Participants who are of Japanese ethnicity (Japanese participant is defined as having both parents and 4 grandparents who are ethnically Japanese and this also includes second and third generation Japanese whose parents or grandparents are living in a country other than Japan)
* Participants who are of Non-Asian ethnicities. A Non-Asian Participant is defined as having both parents and grandparents who are ethnically Non-Asian.
* Body mass index within the range 18 to 32 kg/m^2
* Male and/or female participants of non-child bearing potential

Exclusion Criteria:

* History of any clinically important disease or disorder
* History or presence of gastrointestinal, hepatic, or renal disease or condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Participants with known autoimmune disease or on-treatment with immune-modulatory drugs
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first dose of study intervention
* Any clinically significant cardiovascular event within the last 6 months prior to the Screening Visit
* Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results and any abnormal vital signs
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12-Lead ECG
* Blood dyscrasias with increased risk of bleeding including idiopathic thrombocytopenic purpura and thrombotic thrombocytopenic purpura or symptoms of increased risk of bleeding
* History of major bleed or high-risk of bleeding diathesis
* Participants with a positive diagnostic nucleic acid test for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), at Screening Visit. Participants who test positive for Coronavirus disease 2019 (COVID-19) at Screening Visit
* Participants with a significant COVID-19 illness within 6 months of enrollment
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity
* Received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days of last Follow-up to first dose of study intervention of this study or 5 half-lives from last dose to first dose of study intervention, whichever is the longest
* Participants who have previously received AZD2693
* Previous enrollment or randomization into the present study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Until Day 162 (Final/Early termination visit)
  Safety and tolerability of AZD2693 compared to placebo following multiple dose SC administration in healthy participants will be evaluated.

SECONDARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  Cmax of AZD2693 following single dose SC administration of AZD2693 in healthy participants will be characterized.
Time to reach peak or maximum observed concentration following drug administration (tmax) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  tmax of AZD2693 following single dose SC administration of AZD2693 in healthy participants will be characterized.
Terminal elimination rate constant, estimated by log-linear least-squares regression of the terminal part of the concentration-time curve (λz) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  λz of AZD2693 following single and multiple doses SC administration of AZD2693 in healthy participants will be characterized.
Apparent terminal elimination half-life associated with the terminal slope (λz) of the semi-logarithmic concentration-time curve (t½λz) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  t½λz of AZD2693 following single and multiple doses SC administration of AZD2693 in healthy participants will be characterized. The t½λz , estimated as (ln2)/λz
Area under the plasma concentration-time curve from time zero to 48 hours after dosing AUC (0-48) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  AUC(0-48) of AZD2693 following single and multiple doses SC administration of AZD2693 in healthy participants will be characterized.
Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration (AUClast) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  AUClast of AZD2693 following single and multiple doses SC administration of AZD2693 in healthy participants will be characterized.
Area under the concentration-time curve from time zero extrapolated to infinity. AUCinf is estimated by AUClast + Clast/ λz where Clast is the last observed quantifiable concentration (AUCinf) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  AUCinf of AZD2693 following single dose SC administration of AZD2693 in healthy participants will be characterized.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  CL/F of AZD2693 following single and multiple dose SC administration of AZD2693 in healthy participants will be characterized. CL/F is calculated as Dose/AUCinf for single dose and for multiple dose it is calculated as Dose/AUCτAUCss.
Mean residence time (MRTinf) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  MRTinf of AZD2693 following single dose SC administration of AZD2693 in healthy participants will be characterized.
Time delay between drug administration and the first observed concentration in plasma (tlag) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  tlag of AZD2693 following single and multiple doses SC administration of AZD2693 in healthy participants will be characterized.
Apparent volume of distribution for parent drug at terminal phase (extravascular administration) (Vz/F) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  Vz/F of AZD2693 following single dose SC administration of AZD2693 in healthy participants will be characterized. Vz/F is estimated by dividing the apparent clearance (CL/F) by λz.
Area under the plasma concentration-time curve from time zero to time of last quantifiable analyte concentration divided by the dose administered (AUClast/D) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  AUClast/D of AZD2693 following single and multiple doses SC administration of AZD2693 in healthy participants will be characterized.
Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by the dose administered (AUCinf/D) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  AUCinf/D of AZD2693 following single dose SC administration of AZD2693 in healthy participants will be characterized.
Observed maximum plasma concentration divided by the dose administered (Cmax/D) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  Cmax/D of AZD2693 following single and multiple doses SC administration of AZD2693 in healthy participants will be characterized.
Time of the last quantifiable concentration (tlast) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  tlast of AZD2693 following single and multiple doses SC administration of AZD2693 in healthy participants will be characterized.
Maximum observed plasma drug concentration at steady state (Cmax) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  Cmax of AZD2693 following multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Minimum observed drug concentration at steady state (Cmin) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  Cmin of AZD2693 following multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Time to reach maximum observed plasma concentration at steady state (tmax) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  tmax of AZD2693 following multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Area under the concentration-time curve in the dose interval (AUCτ) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  AUCτ of AZD2693 following multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by the dose administered (AUCτ/D) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  AUCτ/D of AZD2693 following multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Accumulation ratio based on Cmax (Rac Cmax) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  Rac Cmax of AZD2693 following multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Accumulation ratio based on AUC (Rac AUC) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  Rac AUC of AZD2693 following multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Temporal change parameter in systemic exposure (TCP) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose), Day 8, Day 29 (pre-dose only), and days 64, 78, 92, 106, 120, 134, 148, and 162 (Final/ET visit)
  TCP of AZD2693 following multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Amount of analyte excreted into the urine from time t1 to t2 (Ae(t1-t2)) for AZD2693 | Day 1 and Day 57 (pre-dose and post-dose)
  (Ae(t1-t2)) of AZD2693 following single and multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Cumulative amount of analyte excreted from time zero through the last sampling interval Ae(0-last) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose)
  Ae(0-last) of AZD2693 following single and multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Fraction of dose excreted unchanged into the urine from time t1 to t2 fe(t1-t2) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose)
  fe(t1-t2) of AZD2693 following single and multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Cumulative fraction (percentage) of dose excreted unchanged into the urine from time zero to the last measured time point (fe(0-last)) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose)
  fe(0-last) of AZD2693 following single and multiple dose SC administration of AZD2693 in healthy participants will be characterized.
Renal clearance of drug from plasma, estimated by dividing Ae(0-t) by AUC(0-t) where the 0-t interval is the same for both Ae and AUC (CLR) of AZD2693 | Day 1 and Day 57 (pre-dose and post-dose)
  CLR of AZD2693 following single and multiple dose SC administration of AZD2693 in healthy participants will be characterized.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7830C00006&attachmentIdentifier=223dd36e-57ce-40a4-8de7-f8e2d671f7ea&fileName=D7830C00006_Redacted_CSR_synopsis.pdf&versionIdentifier=